CLINICAL TRIAL: NCT01695824
Title: Implantation of Left Atrial Appendage Occluders Concomitantly With Catheter Ablation in Patients With Atrial Fibrillation
Brief Title: Left Atrial Appendage (LAA) Occluders After Catheter Ablation of Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WA-PR-AF
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Atrial Fibrillation
Keywords: catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LAA occluder (Active Comparator)
  Interventions: Device: LAA occluder; Procedure: RFA ablation; Drug: Warfarin
- Warfarin (Active Comparator)
  Interventions: Procedure: RFA ablation; Drug: Warfarin

INTERVENTIONS:
Device: LAA occluder — The procedure is performed under transesophageal echocardiographic (TEE) guidance. After a transseptal puncture is performed, a pigtail catheter is maneuvered into the LAA to perform an LAA angiogram. Through the use of a combination of this angiographic and TEE information, a Watchman device, ranging in size between 21 and 33 mm in diameter, is selected. The device comes prepackaged in a catheter-based delivery system that is advanced into the LAA through a 12F transseptal sheath (outer diameter, 14F). Proper positioning and stability of the device are verified by TEE and angiography before device release.
  Other Names: Watchman
  Arms: LAA occluder
Procedure: RFA ablation — The left atrium (LA) and pulmonary veins (PVs) were explored through a transseptal approach. Real-time three-dimensional (3D) LA maps were reconstructed by using a nonfluoroscopic navigation system (CARTO, Biosense-Webster Inc.). The ipsilateral left and right PVs were encircled in 1 lesion line by circumferential PV isolation. Radiofrequency energy was delivered at 43◦C, 35 W, 0.5 cm away from the PV ostia at the anterior wall, and was reduced to 43◦C, 30 W, 1 cm away from the PV ostia at the posterior wall, with a saline irrigation speed of 17 mL/min. Each lesion was ablated continuously until the local potential amplitude decreased by >80% or RF energy deliveries exceeded 40 seconds. The endpoint of circumferential PV isolation was PV isolation; this was confirmed when Lasso mapping showed the disappearance of all PV potentials or the dissociation of PV potentials from left atrial activity.
Drug: Warfarin — Warfarin was discontinued in 45 days after procedure in case of no trombus by TE for "Watchman group"
  All patients in "Warfarin group" continued to receive Warfarin during hole study period with IMR from II to III.

SUMMARY:
The primary objective of this study is to assess combined end point (All stroke, Systemic embolism, Cardiovascular death) between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient has paroxysmal, persistent or permanent non-valvular atrial fibrillation (AF)
* Eligible for long term warfarin
* CHADS score >= 1 (congestive heart failure [CHF], history of high blood pressure, 75 years of age or older, diabetes, prior stroke or transient ischemic attack [TIA])

Exclusion Criteria:

* Contraindicated for warfarin
* Contraindicated for aspirin or clopidogrel (Plavix)
* CHF Class 4
* Implanted mechanical valve
* Atrial septal or Patent Foramen Ovale (PFO) device
* Platelets < 100,000 or hemoglobin < 10
* Left ventricular ejection fraction (LVEF) < 30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
All stroke | 12 months
Systemic embolism | 12 months
Cardiovascular death | 12 months

SECONDARY OUTCOMES:
Technical success | 45 days
Procedure success | 45 days
30 day major adverse event (MAE) | 30 days
Left atrial appendage (LAA) coverage | 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology
Locations (1):
- State Research Institute of CIrculation Pathology, Novosibirsk, Russia

REFERENCES:
- [Derived] Romanov A, Pokushalov E, Artemenko S, Yakubov A, Stenin I, Kretov E, Krestianinov O, Grazhdankin I, Risteski D, Karaskov A, Steinberg JS. Does left atrial appendage closure improve the success of pulmonary vein isolation? Results of a randomized clinical trial. J Interv Card Electrophysiol. 2015 Oct;44(1):9-16. doi: 10.1007/s10840-015-0030-4. Epub 2015 Jul 2. PMID 26133284
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru